CLINICAL TRIAL: NCT02538497
Title: The Northern Babies Longitudinal Study: Predicting Postpartum Depression and Improving Parent-infant Interaction With The Newborn Behavioral Observation
Brief Title: The Northern Babies Longitudinal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: Public Health Sisters in the Tromsø municipality (Unknown); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/614REK nord
Record Dates: First submitted 2015-08-04; First posted 2015-09-02 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-04

CONDITIONS: Depression, Postpartum
Keywords: NBO; The Newborn Behavioral Observation; postpartum depression; postnatal depression; child development; parent-child interaction
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO plus routine care (Experimental): The Newborn Behavioral Observation
  Interventions: Behavioral: The Newborn Behavioral Observation (NBO); Behavioral: Routine care
- Routine care (Other)
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: The Newborn Behavioral Observation (NBO) — The Newborn Behavioral Observation (NBO) is a flexible parental guidance methodology which takes between 20 and 40 minutes to administer. It consists of 18 neurobehavioral observations which give a profile of the infant´s behavioral repertoire along the dimensions: attentional-interactional, autonomic, motor and state organization.
  The intervention group will receive 3 NBO consultations: 1) Routine care plus the NBO at the hospital within two days post-delivery; 2) Routine home visit plus the NBO by a public health nurse when the infant is 7-10 days old; and 3) NBO at the well-baby clinic when the infant is about 4 weeks old.
  Other Names: NBO
  Arms: NBO plus routine care
Behavioral: Routine care — The control group will receive routine care. Between 7 and 10 days after birth a public health nurse routinely visits the family at home. Six weeks after birth, the mother and the infant visit the well-baby clinic

SUMMARY:
Postpartum depression (PPD) is a prevalent disorder. Studying the factors related to PPD will help to identify families at risk and provide preventive interventions. This can in turn improve the developmental trajectories for the children. Several previous studies have investigated risk factors for PPD. However, few studies have focused on cognitive vulnerability factors. The first aim of the present study is to explore a range of protective and risk factors, including cognitive factors, for PPD, parent-infant interactions and child development. The second aim of the study is to evaluate the effectiveness of The Newborn Behavioral Observation (NBO) as a universal preventive intervention delivered in routine practice. The NBO is a brief relationship-enhancing intervention that may reduce depressive symptomatology in mothers.

DETAILED DESCRIPTION:
Aims

The present study has three broad aims:

1. Examine key pre- and postnatal predictors related to parental functioning: a) parental depression, anxiety, and stress, b) parental reflective functioning in relation to the infant, and c) parent-infant attachment style.
2. Examine key pre- and postnatal predictors related to interaction and developmental problems in the child: a) difficulties in parent-infant interaction in the first 4 months post-delivery, and b) infant's cognitive, communicative and motor development, signs of sustained withdrawal behaviour, and heart-rate variability at 6 months post-delivery.
3. Evaluate the effectiveness of the NBO as a universal preventive intervention delivered in routine practice as compared to standard care, on:

   * Parental outcomes (depressive symptoms, parenting stress, reflective functioning, attachment to the infant),
   * Relational outcomes (emotional availability in parent-child interaction), and
   * Infant outcomes (cognitive, communicative and motor development at 6 months post-delivery, heart-rate variability).

Predictor variables include some well-known vulnerability factors for developing PPD (e.g., depression symptoms in pregnancy, adult attachment style, relationship satisfaction and life stress), but the main focus in the observational part of the research project is on cognitive vulnerability factors such as early maladaptive schemas, repetitive negative thinking, rumination, implicit attitudes and cognitive processing of emotionally valenced infant facial information.

Study design This is a longitudinal observational study with an intervention. The observational part of the study will use a prospective cohort design. The effect of the intervention will be evaluated using a non-randomized cluster controlled design, since neither cluster nor individual randomization is feasible in this routine practice setting. An intervention group receiving NBO (families belonging to two well-baby clinics in Tromsø municipality) will be compared with a control group (families at the remaining four well-baby clinics in Tromsø) receiving care as usual.

Recruitment All pregnant women and expecting fathers who speak Norwegian are eligible for inclusion in the study. Between autumn 2015 and autumn 2018 approximately 200 families will be recruited by midwifes and by general practitioners (GPs) in the municipality of Tromsø, which is the 9th largest municipality in Norway (~73000 inhabitants; 78). There are approximately 1000 births a year in Tromsø municipality. Based on the experiences from a comparable study, "Little in Norway" (79), the recruitment of 200 families within the project period is considered feasible.

The participants will be recruited in (approximately) week 16 of gestation. At recruitment, women will be given written information about the study and a flyer with an inquiry to be contacted by the research team. If the child's father is not present, the mother is encouraged to inform him about the study. The health worker informs the research team who contacts the women to plan a meeting with them and their partners, preferable between week 16 and 22 of gestation. In this meeting, the prospective parents are given detailed information about the study and are invited to sign an informed consent to participate. In addition, at 4 months post-delivery the parents will be asked to sign an informed consent to obtain birth related information from the birth record.

Power calculations/statistical analysis The sample size is calculated on the basis of differences between intervention group and standard care group on the Edinburgh Postnatal Depression Scale (EPDS) maternal score, the Parenting Stress Index (PSI-PD), the Parental Reflective Functioning Scale (PRFQ) and the Maternal Postnatal Attachment Scale (MPAS) 6 weeks post-delivery. Based on the pilotstudy by Nugent et al. (69) and some regression to the mean, we expect a small to medium effect size (f2 = .07). A MANOVA with the four aforementioned outcome variables can detect a difference between the groups with a power of .80 given a group sizes of N = 176. With an estimated dropout of 10 %, a group size of 200 will be recruited. The estimation is based on an α-level of .05.

Procedure For the observational part of the study, assessments will be performed at six time points (see Table 1): During gestational week 16 - 22 (Step 1), 24 - 30 (Step 2) and 31 (Step 3), and at 6 weeks (Step 4), 4 months (Step 5) and 6 months (Step 6) post-delivery. For the intervention study, pre-intervention measures will be collected at Step 3, post-intervention measures at Step 4 and follow-up measures at Step 5 and 6. Since the families will receive the first NBO already two-days post-delivery, no pre-test assessment can be obtained for the interaction and infant measures. Hence, analyses of intervention effects will be based on differences between groups at 4 and 6 months post-delivery controlling for relevant covariates. The data is collected using online questionnaires, computerized cognitive tests, video-filmed observations of mother-infant interactions, and a standardised test of the child's cognitive, communicative and motor development (Bayley Scales of Infant and Toddler Development; 80).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman and expecting fathers
* Speak Norwegian

Exclusion Criteria:

* Do not speak Norwegian

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Levels of postpartum depression | Six weeks postpartum
  Mothers and fathers self-reported levels of postpartum depression measured with the Edinburgh Postnatal Depression Scale.

SECONDARY OUTCOMES:
Levels of postpartum depression | Four months postpartum
  Mothers and fathers self-reported levels of postpartum depression measured with the Edinburgh Postnatal Depression Scale.
Levels of postpartum depression | Six months postpartum
  Mothers and fathers self-reported levels of postpartum depression measured with the Edinburgh Postnatal Depression Scale.
Parental reflective functioning | Six weeks postpartum
  Mothers and fathers self-reported parental reflective functioning measured with the Parental Reflective Functioning Questionnaire.
Parental reflective functioning | Four months postpartum
  Mothers and fathers self-reported parental reflective functioning measured with the Parental Reflective Functioning Questionnaire.
Bonding between parent and child | Six weeks postpartum
  Self-reported quality of bonding between parent and child measured with Maternal Postnatal Attachment Scale/Paternal Postnatal Attachment Scale.
Bonding between parent and child | Four months postpartum
  Self-reported quality of bonding between parent and child measured with Maternal Postnatal Attachment Scale/Paternal Postnatal Attachment Scale.
Parent-child interaction | Four months postpartum
  Parent-child interaction will be rated on the basis of 15-30 minutes videotaped episodes of parent-infant play interaction.
Parental stress | Six weeks postpartum
  Self-reported measure of parental stress.
Parental stress | Four months postpartum
  Self-reported measure of parental stress.
A composite measure of the infant´s temperament | Six months postpartum
  Parents report of infant´s sensitivity, general activity, frustration tolerance, adaptability, regularity, and soothability.
Infants social withdrawal behaviour | Six months postpartum
  Assessment of the infant's social withdrawal behaviour with The Alarm Distress Baby Scale.
Infant cognitive, communicative and motor development | Six months postpartum
  Assessment of the infant's cognitive, communicative and motor development with The screening test version of Bayley Scales of Infant and Toddler Development
Heart rate variability | Six months postpartum
  Mothers and infants heart rate variability will be measured with a wireless and unobtrusive electrocardiogram (ECG) equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Catharina EA Wang, Professor, Principal Investigator — UiT The Arctic University of Norway
Locations (1):
- UiT The Arctic University of Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hoifodt RS, Nordahl D, Landsem IP, Csifcsak G, Bohne A, Pfuhl G, Rognmo K, Braarud HC, Goksoyr A, Moe V, Slinning K, Wang CEA. Newborn Behavioral Observation, maternal stress, depressive symptoms and the mother-infant relationship: results from the Northern Babies Longitudinal Study (NorBaby). BMC Psychiatry. 2020 Jun 15;20(1):300. doi: 10.1186/s12888-020-02669-y. PMID 32539729
- [Derived] Hoifodt RS, Nordahl D, Pfuhl G, Landsem IP, Thimm JC, Ilstad LKK, Wang CEA. Protocol for the Northern babies longitudinal study: predicting postpartum depression and improving parent-infant interaction with The Newborn Behavioral Observation. BMJ Open. 2017 Sep 27;7(9):e016005. doi: 10.1136/bmjopen-2017-016005. PMID 28963284